CLINICAL TRIAL: NCT02506335
Title: Liver Function Measured by HepQuant-SHUNT in the Prediction of Outcomes in Patients With Passive Hepatic Congestion Secondary to Congenital Heart Disease (CHD) or Cardiomyopathy
Brief Title: Liver Function Measured by HepQuant-SHUNT in the Prediction of Outcomes in Patients With Heart Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Daniel Ganger, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00100794
Record Dates: First submitted 2015-06-24; First posted 2015-07-23 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Liver Disease; Cardiovascular Disease
Keywords: Liver disease; cardiomyopathy; congenital heart disease
MeSH Terms: conditions — Liver Diseases; Cardiovascular Diseases; Cardiomyopathies; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hep quant cholate testing (Other): diagnostic measure of liver function
  Interventions: Drug: Cholate testing

INTERVENTIONS:
Drug: Cholate testing — The patient receives simultaneously an oral dose of d4-cholate and an IV dose of 13C-cholate, which are stable isotopes; there is no radioactivity or radiation exposure.
  Other Names: 13C-cholate; d4-cholate

SUMMARY:
Background: It is still difficult to predict the outcome in patients requiring Fontan Revisions and in those who have evidence of congestive hepatopathy and probable cirrhosis requiring major cardiac surgery including heart transplant. Over the years, many prognostic indices have been derived from laboratory results of blood tests, clinical and physiological variables (or some combination thereof), from liver imaging to liver histology, which has issues of sampling error, medical risks and technical difficulty. None of these have proved entirely satisfactory. Predicting morbidity or survival is particularly important when deciding about Fontan revisions versus the need for heart transplantation. What is needed here is a truly reliable test of liver function that can help predict outcome, on the basis of a single measurement within few days of a planned revision. For this purpose, it is desirable that the chosen tests of liver performance be safe, non-invasive, easy to perform, have a rapid turnaround for results, and be readily repeatable.

Tests of hepatic elimination of various exogenous substances have been described, such as galactose elimination capacity (GEC), indocyanine green (ICG) clearance, lidocaine metabolism to monoethylglycinexylidide (MEGX), and other tests that rely on liver metabolic capacity. None of these metabolic or clearance tests achieved widespread acceptance or use, mostly because their performance and analyses were cumbersome.

HepQuant,LLC has developed a platform of tests of liver function which include Systemic Hepatic Filtration Rate (HFR), Portal HFR, SHUNT, and Disease Severity Index (DSI)1,2. HepQuant tests specifically target the hepatic uptake of cholate and use a single noninvasive test of 90 minutes duration to quantify the systemic circulation, portal circulation, and portal-systemic shunt and to derive a DSI in intact human subjects. HepQuant tests can assess all stages and etiologies of liver disease. In chronic HCV patients HepQuant testing can predict which patients will respond to antiviral therapy and can measure the improvement in hepatic function that occurs after successful antiviral therapy. Patients who did not respond were followed for an average of 5 years and up to 8 years, and baseline HepQuant testing could predict clinical outcomes (CTP progression, variceal bleeding, encephalopathy, ascites, liver-related death) with 87% sensitivity and 71% specificity.

DETAILED DESCRIPTION:
Hypothesis The results of HepQuant in patients with CHD will correlate with outcomes of cardiac surgery (namely morbidity as defined by complications such as ischemic hepatitis, survival, need for heart transplantation, improvement of liver function post revision), and thus can be used for prognosis in this condition, either alone or in conjunction with other clinical, physiological, and laboratory prognostic scores, thereby giving clinical guidance concerning the need for heart transplantation and simultaneous liver transplantation..

Primary Aim To assess the relationship between HepQuant testing results and clinical outcomes in patients with liver disease secondary to congenital heart disease (CHD) undergoing Fontan revisions.

To assess the clinical outcomes of patients with liver disease secondary to acquired cardiomyopathy or valvular disease that will undergo extensive heart surgery or heart transplantation.

Secondary Aim To assess whether HepQuant testing predicts clinical outcome in patients with Liver Disease and CHD when used in conjunction with other diagnostic tests, such as MELD, Child-Turcotte-Pugh (CTP), liver stiffness measurement (US with ARFI), and Fibrotest (Fibrosure).

Study population Male and female Subjects (age 18 to 70 years) with liver disease secondary to congenital heart disease or cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-specific assessments.
2. Liver disease secondary to congenital heart disease or cardiomyopathy.
3. Male and female subjects (age 18 to 70 years of age).

Exclusion Criteria:

1. Male and female subjects < 18 or > 70 years of age.
2. Female subjects of child-bearing potential that are pregnant or breast feeding.
3. Subjects on both beta blockers and ACE inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Liver Function | 6 months
  Liver function as measured by HepQuant testing which include Systemic Hepatic Filtration Rate (HFR), Portal HFR, SHUNT.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ganger, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Everson GT, Shiffman ML, Morgan TR, Hoefs JC, Sterling RK, Wagner DA, Kulig CC, Curto TM, Wright EC; Halt-C Trial Group. The spectrum of hepatic functional impairment in compensated chronic hepatitis C: results from the Hepatitis C Anti-viral Long-term Treatment against Cirrhosis Trial. Aliment Pharmacol Ther. 2008 May;27(9):798-809. doi: 10.1111/j.1365-2036.2008.03639.x. Epub 2008 Feb 7. PMID 18266997
- [Result] Everson GT, Martucci MA, Shiffman ML, Sterling RK, Morgan TR, Hoefs JC; HALT-C trial group. Portal-systemic shunting in patients with fibrosis or cirrhosis due to chronic hepatitis C: the minimal model for measuring cholate clearances and shunt. Aliment Pharmacol Ther. 2007 Aug 1;26(3):401-10. doi: 10.1111/j.1365-2036.2007.03389.x. PMID 17635375

DOCUMENTS (1):
  • Informed Consent Form (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02506335/ICF_000.pdf